CLINICAL TRIAL: NCT00152802
Title: Immunogenicity of Pneumococcal Vaccine in Liver Transplant Recipients Using a Conjugate-Polysaccharide Priming-Booster Strategy
Brief Title: Pneumonia Vaccine in Liver Transplant Recipients: a Booster Strategy Using a Conjugate Vaccine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Health Network, Toronto (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 04-0450-A
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Last update posted 2007-02-19 (Estimated); Status verified 2005-09

CONDITIONS: Transplant
Keywords: liver transplant; antibody response; opsonophagocytic assay; pneumococcal conjugate vaccine; pneumococcal polysaccharide vaccine

INTERVENTIONS:
Biological: The polysaccharide vaccine Pneumovax (Merck-Frosst)
Biological: The conjugate vaccine used will be Prevnar (Wyeth vaccines)

SUMMARY:
The trial will compare a group of patients whose immune system is primed with the pneumococcal conjugate vaccine and then given a boost with polysaccharide vaccine (prime-boost strategy) vs. a group vaccinated with the standard 23-valent polysaccharide vaccine alone. It is hypothesized that the conjugate vaccine priming will provide an enhanced response in these immunosuppressed individuals who may respond poorly to standard vaccination.

DETAILED DESCRIPTION:
OBJECTIVE: Responses to 23-valent polysaccharide pneumococcal vaccine (PPV23) are poor in organ transplant recipients. We have recently shown that the conjugate pneumococcal vaccine (PCV7) is immunogenic in this population but responses remain suboptimal. This is a clinical study designed to assess the immunogenicity of a novel pneumococcal vaccination strategy in a cohort of adult liver transplant recipients. The trial will compare a group of patients primed with the pneumococcal conjugate vaccine plus polysaccharide boost with a group primed with placebo plus the standard 23-valent polysaccharide vaccine.

Specific objectives of this study are:

* To determine the quantitative antibody response using both vaccine strategies
* To determine the functional antibody response by the opsonophagocytic assay. This assay has the advantage of assessing if patient antibody responses represent truly functional antibodies that display opsonic activity against pneumococcus and is likely better correlated with protective efficacy.
* To determine the durability of response over two years In addition, the safety of the conjugate vaccine and a determination of whether time from transplant affects response to vaccination will be made.

HYPOTHESIS: It is hypothesized that the PCV7 priming will provide an enhanced response in these immunosuppressed individuals who may respond poorly to standard vaccination.

RESEARCH PLAN: We will enroll 130 liver transplant recipients from the out-patient transplant clinics at Toronto General Hospital, Toronto, Ontario. Recipients who have had pneumococcal vaccination in the past 5 years will be excluded. Upon enrolment, patients will be randomized to receive either placebo or PCV7 in a blinded fashion. Eight weeks later, all subjects will receive PPV23. Serum will be obtained at baseline, 8 weeks, 16 weeks, 6, 12, 18, and 24 months. Sera will be used to perform antibody testing to seven pneumococcal serotypes (4, 6B, 9V, 14, 18C, 19F, 23F). The baseline, 8, and 16 week sera will be used for opsonophagocytic assay to the above seven serotypes. A baseline nasopharyngeal swab will also be obtained to look for colonization with Streptococcus pneumoniae. Patient recruitment is expected to take two years and follow-up of all patients should be complete by year 3. An additional 4 months will be needed to complete all laboratory testing. The primary outcome will be anticapsular antibody concentration at 16 weeks. A serotype response will be defined as a 2-fold or greater rise in titer from the 8 week concentration. A vaccine response will be defined as response to at least one serotype of the seven measured.

FUTURE DIRECTIONS: Results of this trial will help to develop a rational and optimal pneumococcal vaccination strategy that would prevent significant morbidity in organ transplant recipients. We are currently studying the impact of pneumococcal disease in transplantation by: (i) a review of invasive pneumococcal disease in transplant recipients in Toronto-Peel region to determine incidence and predominating serotypes; (ii) a Canadian survey of vaccination practices in transplantation; (iii) a 3-year follow-up study to determine the sustainability of immune response to pneumococcal vaccine in renal transplant patients previously enrolled in a vaccine trial. We hope that these studies will form the basis of pneumococcal vaccination recommendations for organ transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

Male or female outpatients who fulfill the following criteria will be eligible for the study:

* Liver transplant recipients greater than 3 months post-transplant
* No prior pneumococcal vaccination within the last 5 years
* Stable allograft function as evidenced by a alanine aminotransferase <10 times the upper limit of normal (mmol/L) that is not worsening
* Able to provide written informed consent and comply with study protocol
* Age > 16

Exclusion Criteria:

* Unable to provide informed consent or comply with protocol
* Prior pneumococcal vaccination within 5 years of enrolment
* Splenectomy
* Admitted to hospital for acute illness
* Febrile illness in the past 2 weeks
* Intravenous Immunoglobulin in the last 6 months
* Current episode of allograft rejection
* Currently on full-dose anticoagulation as a contraindication to intramuscular injection

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130
Dates: Start 2005-01; Study Completion 2009-01

PRIMARY OUTCOMES:
Antibody titres to the seven serotypes contained in conjugate vaccine (4, 6B, 9V, 14, 19F, 23F) measured at baseline, 8 and 16 weeks. Primary outcome measure will be the anticapsular antibody concentration at 16 weeks.

SECONDARY OUTCOMES:
i) Functional Antibody concentration: The titer of functional antibody against the seven pneumococcal serotypes contained in the conjugate vaccine will be determined
ii) Adverse Reactions: Any adverse effects attributed to conjugate or polysaccharide vaccines will be documented. These will include local reactions such as redness, swelling, tenderness and systemic reactions such as fever.
iii) Invasive Pneumococcal Disease: The study is not sufficiently powered to look at differences in pneumococcal disease between the two groups. However, any occurrence of documented pneumococcal disease in vaccinated patients will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Deepali Kumar, BSc, MSc, MD, FRCP(C), Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Kumar D, Chen MH, Wong G, Cobos I, Welsh B, Siegal D, Humar A. A randomized, double-blind, placebo-controlled trial to evaluate the prime-boost strategy for pneumococcal vaccination in adult liver transplant recipients. Clin Infect Dis. 2008 Oct 1;47(7):885-92. doi: 10.1086/591537. PMID 18715160